CLINICAL TRIAL: NCT00322790
Title: INST 0549C Differences in 30-year Trends in Incidence and Survival for Malignant Germ Cell Tumors in Males and Females: A SEER Population-based Study
Brief Title: Differences in Trends Malignant Germ Cell Tumors in Males and Females: A SEER Population-based Study
Status: Withdrawn | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0549C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Differences in 30-year Trends in Incidence and Survival for Malignant Germ Cell Tumors in Males and Females.

DETAILED DESCRIPTION:
Differences in 30-year Trends in Incidence and Survival for Malignant Germ Cell Tumors in Males and Females: A SEER Population-based Study.

ELIGIBILITY:
Inclusion Criteria:

* Survival for Malignant Germ Cell Tumors in Males and Females.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with malignant germ cell tumors at University of New Mexico facilities
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Estimated); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States